CLINICAL TRIAL: NCT03074591
Title: Effect of IV Iron (Ferric Carboxymaltose, Ferinject) on Exercise Tolerance, Symptoms and Quality of Life in Patients With Heart Failure With Preserved Ejection Fraction (HFpEF) and Iron Deficiency With and Without Anaemia.
Brief Title: Effect of IV Iron in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: FAIR-HFpEF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Göttingen (Other)
Responsible Party: Principal Investigator, Prof. Stefan D Anker, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Charite
Record Dates: First submitted 2017-03-01; First posted 2017-03-09 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Iron-deficiency; Heart Failure
Keywords: Iron deficiency; Heart failure
MeSH Terms: conditions — Anemia, Iron-Deficiency; Heart Failure; Iron Deficiencies | interventions — ferric carboxymaltose; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Active treatment: Ferric Carboxymaltose solution (Ferinject®) for parenteral application, 50 mg/mL iron. Medication will be given as a short time infusion over 15 minutes in 100mL NaCl.
  Interventions: Drug: Ferric Carboxymaltose 50Mg/Ml Inj 15Ml
- Placebo (Placebo Comparator): Placebo: Normal saline (0.9% weight/volume (w/v) NaCl) administered in analogy to active treatment procedures.
  Interventions: Drug: Saline Solution for Injection

INTERVENTIONS:
Drug: Ferric Carboxymaltose 50Mg/Ml Inj 15Ml — After baseline assessments patients will be randomised in a 1:1 ratio to receive Ferric Carboxymaltose IV or placebo/saline (normal saline: 0.9% w/v NaCl). In the Treatment group, Ferric Carboxymaltose will be administered according to the dosing schedule.
  Other Names: Ferric Carboxymaltose
  Arms: Treatment
Drug: Saline Solution for Injection — In the placebo/saline group, patients will receive the aequivalent number of normal saline infusions.
  Other Names: Saline Solution
  Arms: Placebo

SUMMARY:
This study addresses, whether treatment with IV iron for patients with heart failure with preserved ejection fraction (HFpEF) and iron deficiency (ID), both with or without anaemia, can improve exercise capacity as measured by 6-minute walking test (6-MWT) and symptoms while being safe

DETAILED DESCRIPTION:
All previous trials have excluded patients with HFpEF. This study addresses, whether treatment with IV iron for patients with heart failure with preserved ejection fraction (HFpEF) and iron deficiency (ID), both with or without anaemia, can improve exercise capacity as measured by 6-minute walking test (6-MWT) and symptoms while being safe. The FAIR-HFpEF study was designed to evaluate the efficacy of Ferinject® in improving symptoms of HFpEF in patients with ID. Analyses will focus both on subjective and objective measures as well as on patients with and without anaemia. Furthermore, the tolerability and safety of Ferinject® treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing to participate and provides written informed consent;
2. Age ≥18 years;
3. Clinical diagnosis of heart failure with preserved ejection fraction (HFpEF) with LVEF ≥45% at screening or within 6 months prior to planned randomisation (assessed by echocardiography or MRI);
4. Ambulatory for at least 7 days with NYHA class II or III at time of randomisation (the screening visit can take place at the end of a hospitalisation);
5. Treated with a diuretic;
6. Presence of atrial fibrillation (AF) at screening or randomisation is allowed in 2 out of 4 patients (calculated per centre);
7. At screening or randomisation, presence of one of the following criteria:

   1. hospitalisation with a diagnosis of HF within 12 months prior to planned randomisation; OR
   2. raised plasma levels of natriuretic peptides in a patient with sinus rhythm (i.e. in patients without AF: NT-proBNP >300 pg/mL or BNP >100 pg/mL or MR-proANP >120 pmol/L; in patients with AF: NT-proBNP >600 pg/mL or BNP >200 pg/mL or MR-proANP >250 pmol/l)
8. Evidence of diastolic dysfunction at screening or randomisation, defined as:

   1. E/E' >13; OR
   2. LA width ≥38 mm; OR
   3. LA length ≥50 mm; OR
   4. LA area ≥20 cm2; OR
   5. LA volume ≥55 ml; OR
   6. left atrial volume index >28 mL/m2;
9. Haemoglobin >9.0 g/dL and ≤14.0 g/dL (at screening);
10. ID with ferritin <100 ng/mL or ferritin 100-299 plus TSAT <20% (at screening);
11. 6-minute-walking distance at baseline <450 m (average of the last 2 documented tests within 8 weeks prior to planned randomisation that also need to be within 20% of each other).

Exclusion Criteria:

1. Unable to sign informed consent
2. Any prior echocardiography measurement of LVEF <40%;
3. Clinical signs and symptoms of infection including fever >38°C;
4. Use of IV iron, erythropoietin or blood transfusions within the previous 60 days;
5. Use of concurrent immunosuppressive therapy;
6. History of acquired iron overload or haemochromatosis (or a first relative with haemochromatosis);
7. Known hypersensitivity to FCM or any other IV iron product;
8. Known bleeding or haemolytic anemia;
9. Presence of any condition that precludes exercise testing, such as decompensated HF, significant musculoskeletal disease, unstable angina pectoris, obstructive cardiomyopathy, severe uncorrected valvular disease, or uncontrolled brady-arrhythmias or tachy-arrhythmias;
10. Probable alternative diagnoses that in the opiniton of the investigator could account for the patient's HF symptoms such as severe obesity, primary pulmonary hypertension, or chronic obstructive pulmonary disease (COPD); hence, patients with the following are excluded:

    1. Severe COPD, i.e. with known FEV1 <50%, requiring home oxygen therapy, or on chronic oral steroid therapy;
    2. body mass index ≥40.0 kg/m2;
11. Presence of uncontrolled atrial fibrillation with resting heart rate >110/min;
12. Presence of uncontrolled hypertension with blood pressure >160/100 mm Hg;
13. Renal replacement therapy;
14. Concurrent therapy with an erythropoiesis stimulating agent;
15. Known active malignancy;
16. Known HIV or active hepatitis infection;
17. Pregnancy;
18. Patients, who may be dependent on the sponsor, the investigator or the trial sites, have to be excluded from the trial
19. Lack of willingness to storage and disclosure of pseudonymous disease data in the context of the clinical trial.
20. Participation in another clinical trial within previous 30 days and/ or anticipated participation in another trial during this study.
21. Inability to fully comprehend and/or perform study procedures in the investigator's opinion;
22. Persons staying at an institution due to order by a national body or a court of law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
exercise capacity | 24 weeks
  The difference of 6-minute walking distance in meters from baseline to week 24 in symptomatic patients with HFpEF with documented ID compared to the control group.

SECONDARY OUTCOMES:
6min-walking distance | 52 weeks
  Difference in 6-minute walking distance in meters from baseline to end of study in symptomatic patients with HFpEF with documented ID compared to the control group
Patient Global Assessment (PGA) | 52 weeks
  Difference in Patient Global Assessment (PGA) in symptomatic patients with HFpEF with documented ID from baseline to end of study.
  (7-point Likert scale [non-parametric])
NYHA functional class | 52 weeks
  Difference in NYHA class from baseline to end of study in symptomatic patients with HFpEF
Change in quality of life assessments | 52 weeks
  Difference in quality of life assessments (EQ-5D (= European Quality of Life 5 Dimensions 3 Level Version; = tool for Patient-Reported Outcomes (PRO) measurement); KCCQ (= Kansas City Cardiomyopathy Questionnaire)) from baseline to end of study in symptomatic patients with HFpEF.
  KCCQ: (0-100) -> 100=best
  EQ-5D (5-point Likert scale, 5 dimensions (mobility, self-care, usual activities, pain, anxiety) 5 levels (1 = no problems level 5 = extreme problems))
Rate of recurrent heart failure hospitalisations and death | 52 weeks
  Difference in the rate of recurrent heart failure hospitalisations and deaths in symptomatic patients with HFpEF and ID.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Anker, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (7):
- Germany (7):
  - Innere Medizin/Kardiologie, Nuremberg, Bavaria
  - University Medical Center Göttingen, Göttingen, Lower Saxony
  - Saarland University Medical Center, Homburg, Saarland
  - Herzzentrum Dresden GmbH, Dresden, Saxony
  - Charité University Medicine Berlin, Berlin
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Herzklinik Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication of main results

REFERENCES:
- [Background] von Haehling S, Doehner W, Evertz R, Garfias-Veitl T, Diek M, Karakas M, Birkemeyer R, Fillippatos G, Ponikowski P, Böhm M, Friede T, Anker SD. Iron deficiency in heart failure with preserved ejecton fracton: ratonale and design of the FAIR-HFpEF trial. Global Cardiol 2023; 1: 39-46.
- See also: Related Info — https://www.globalcardiology.info/site/article/view/15